CLINICAL TRIAL: NCT03842514
Title: Investigation of the Effects of Dietary Lecithin on Intestinal Permeability, Bacterial Translocation, Microbiota and Glucose Metabolism
Brief Title: Food Additives - Do Processed Diets Impact on Gut and Metabolic Health
Acronym: FADiets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: Medical Research Council (Other Government); University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 810
Record Dates: First submitted 2019-02-06; First posted 2019-02-15 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Gut Health; Metabolic Health
MeSH Terms: interventions — bearberry, bladderwrack, borage oil, centella, fatty acid, fish oil, ginkgo biloba, melilotus, soya lecithin drug combination

STUDY DESIGN:
Intervention Model Description: Diet trial with randomised sequence of delivery of two diets.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-emulsifier to Low-emulsifier (Experimental): Phase 1: No intervention - 7 days food diary (recording at home, usual diet)
  Phase 2: 14 days high-emulsifier (soya lecithin) low-calorie diet at 100% resting metabolic rate
  Phase 3: No intervention - 7 days washout with usual diet
  Phase 4: 14 days low-emulsifier low-calorie diet at 100% resting metabolic rate
  Interventions: Dietary Supplement: Soya lecithin
- Low-emulsifier to High-emulsifier (Experimental): Phase 1: No intervention - 7 days food diary (recording at home, usual diet)
  Phase 2: 14 days low-emulsifier low-calorie diet at 100% resting metabolic rate
  Phase 3: No intervention - 7 days washout with usual diet
  Phase 4: 14 days high-emulsifier( soya lecithin) low-calorie diet at 100% resting metabolic rate
  Interventions: Dietary Supplement: Soya lecithin

INTERVENTIONS:
Dietary Supplement: Soya lecithin — The lecithin supplement will be soya lecithin granules given as 7.5 g twice daily, incorporated into juices

SUMMARY:
This dietary intervention study will assess the effect in healthy human volunteers of an E number which is a food additive and commonly used and consumed emulsifier, on gut function, gut inflammation and glucose metabolism. We will be using a powdered soy lecithin product in the food to compare a diet with and without this ingredient.

DETAILED DESCRIPTION:
A dietary intervention study to investigate the effect, in healthy human volunteers, of dietary lecithin (soy lecithin), a commonly used/consumed emulsifier, on markers of gut function particularly bacterial translocation (assessed by measure of venous blood bacterial DNA, circulating lipopolysaccharide [LPS] binding protein and soluble CD14), gut inflammation (assessed by measurement of faecal calprotectin), gut microbiota activity/composition (faecal short-chain fatty acid [SCFA] profile and bacterial diversity [16S ribosomal RNA genes]) and glucose metabolism (measured by oral glucose tolerance test [OGGT], plasma fasted lipids and insulin).

ELIGIBILITY:
Inclusion Criteria:

• BMI ranging from 27-40 kg/m2

Exclusion Criteria:

* Antibiotic use within the past 3 months (due to impact on gut microbiota)
* Current Statin use
* Current Aspirin use
* Chronic inflammatory disorders (including rheumatoid arthritis, inflammatory bowel disease)
* Food allergies or self-reported food sensitivity or intolerance
* Diagnosis of diabetes
* Pregnant or breastfeeding
* Unsuitable veins for blood sampling
* Inability to speak, read and understand English
* Unable to comply to alcohol-free diet for 5 weeks
* Consumption of nutrition supplements
* Soy allergy or intolerance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Change in bacterial translocation | Samples collected at baseline and after each 14 day intervention period. Will be assessed no later than 48 months post final volunteer completion
  Assessment of change in bacterial translocation by venous blood bacterial DNA measured as responding to pre and post dietary treatment as gene copy number per ml but using more validated universal qPCR primer sets (including total bacteria, phyla- and class-specific primers)

SECONDARY OUTCOMES:
Faecal calprotectin | Samples collected at baseline and after each 14 day intervention period. Will be assessed no later than 48 months post final volunteer completion
Faecal volatile organics compounds | Samples collected at baseline and after each 14 day intervention period. Will be assessed no later than 48 months post final volunteer completion
Faecal short chain fatty acids | Samples collected at baseline and after each 14 day intervention period. Will be assessed no later than 48 months post final volunteer completion
Faecal bacterial 16S rRNA gene sequencing | Samples collected at baseline and after each 14 day intervention period. Will be assessed no later than 48 months post final volunteer completion
Plasma highly sensitive C-reactive protein | Samples collected at baseline and after each 14 day intervention period. Will be assessed no later than 48 months post final volunteer completion
Plasma soluble CD14 and LPS binding protein | Samples collected at baseline and after each 14 day intervention period. Will be assessed no later than 48 months post final volunteer completion
Plasma fasting blood glucose and up to 3 hours after OGTT | Samples collected at baseline and after each 14 day intervention period. Will be assessed no later than 48 months post final volunteer completion
Plasma fasted insulin profile and up to 2 hours postprandial OGTT | Samples collected at baseline and after each 14 day intervention period. Will be assessed no later than 48 months post final volunteer completion
Plasma fasting lipid profile | Samples collected at baseline and after each 14 day intervention period. Will be assessed no later than 48 months post final volunteer completion
  Triglycerides, high and low-density cholesterol will be assessed by Kone automated analyser
Plasma trimethylamine-N-oxide (TMAO) | Samples collected at baseline and after each 14 day intervention period. Will be assessed no later than 48 months post final volunteer completion

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Johnstone, PhD, Principal Investigator — University of Aberdeen
Locations (1):
- The Rowett Institute, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-18): https://cdn.clinicaltrials.gov/large-docs/14/NCT03842514/Prot_SAP_001.pdf